CLINICAL TRIAL: NCT05428163
Title: Immunophenotyping of Plasma Cells and Immune Effector Cells in Peripheral Whole Blood and Bone Marrow Samples From Multiple Myeloma (MM) Patients
Acronym: MYELOME-MM
Status: Completed | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: RCAPHM20_0012 - MYELOME-MM; 2020-A01783-36 (Other: ANSM)
Record Dates: First submitted 2022-06-14; First posted 2022-06-22 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Multiple Myeloma
Keywords: Immune response; Plasma cells; Multiple myeloma; Drugs targeting plasma cells
MeSH Terms: conditions — Multiple Myeloma | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Biological sampling — 3ml of blood
  Other Names: blood sampling

SUMMARY:
The objective of this study is to evaluate the immune profile of plasma cells and immune effector cells in paired peripheral whole blood and bone marrow samples from MM patients by standardized flow cytometry. The quantitative and/or qualitative variation of these immune effectors according to the different status of myeloma pathology (diagnosis, relapse or refractory). It is interesting to assess the extent to which a particular immune profile is associated with a better therapeutic response for a given treatment.

In addition, the study will validate the stability of the samples between T0 (< 4 hours after sampling) and T0 + 72 hours.

DETAILED DESCRIPTION:
Study the biomarkers recorded on plasma cells and normal leukocytes including T lymphocytes (naïve, effectors and memories), B lymphocytes, Treg, NK, monocytes as well as their activation markers (CD25, PD-1) in paired bone marrow and blood samples. Validate the pre-analytical stability of the samples between T0 (< 4 hours after sampling) and T0 + 72 hours.

Secondary objectives: Validate the strategy of quantification of receptors on plasma cells by direct labeling in flow cytometry. Validate a new method for measuring receptor occupancy by a drug. Validate the pre-analytical stability of the absolute quantitative expression of the receptors and the specific marker CD138 on samples between T0 (< 4 hours after sampling) and T0 + 72 hours.

The study will be enrolling 20 patients.

ELIGIBILITY:
Inclusion Criteria:

* Multiple myeloma without treatment

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with Multiple myeloma without treatment
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-10-04 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
immunophenotyped cells | day 0; day0+24hour; day 0+ 48hours; day0+72hours
  change in % of immunophenotyped cells during time

CONTACTS AND LOCATIONS:
Overall Officials: Regis Costello, Principal Investigator — AP-HM
Locations (1):
- APHM, Marseille, France

IPD SHARING:
Plan to Share IPD: No